CLINICAL TRIAL: NCT02678806
Title: Radiotherapy in Hepatocellular Carcinomas After Hepatectomy With Narrow Margin (<1 cm) and / or Microvascular Invasion
Acronym: RHCC:BCLC-A
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangxi Medical University (Other)
Responsible Party: Principal Investigator, TaoBai, Researcher, Guangxi Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GDWTaoBai
Record Dates: First submitted 2016-01-23; First posted 2016-02-10 (Estimated); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: HepatoCellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Postoperative radiotherapy group (Experimental): Patients hospitalized in Affiliated Tumor Hospital of Guangxi Medical University from 1st November 2017, who were diagnosed as BCLC-A stage hepatocellular carcinoma, accepted hepatocellular carcinoma resection, pathologically confirmed as narrow margin (the closest distance from margin to tumor capsule < 1cm) and microvascular invasion was found in tumor capsule and adjacent tissues junction were selected and received margin postoperative radiotherapy.
  Interventions: Radiation: Postoperative radiotherapy
- Postoperative TACE group (Active Comparator)
  Interventions: Drug: Postoperative TACE

INTERVENTIONS:
Radiation: Postoperative radiotherapy — The radiotherapy group received prophylactic radiotherapy 1 month after operation. All the patients in the experimental group were treated with 6 to 8 MV X-ray, intensity-modulated irradiation (IMRT) technique, which was divided into 4-5 fields, 2Gy/25 times. 5f/W, total dose 50Gy
  Arms: Postoperative radiotherapy group
Drug: Postoperative TACE — In the intervention group, TACE was performed in January and March after operation. The femoral artery puncture was performed by Seldinger method, and the cannula was intubated to the hepatic artery by DSA. Then, 50 mg of lobaplatin plus 4 mg of raltitrexed was injected into the vascular artery. The embolic agent was selected as 38.0. % super liquefied iodine solution and / or gelatin sponge particles, the dose is maintained at 5 ~ 20ml. At the end of treatment, a DSA examination again confirmed that the tumor was completely occluded.
  Arms: Postoperative TACE group

SUMMARY:
Hepatocellular carcinoma is one of ten leading cancer types worldwide and also in Asia, but the five-year relative survival rate is relatively quite low1-3. For hepatocellular carcinoma treatment, current options are surgical resection, embolization chemotherapy, radiation therapy, a variety of ablation therapy, biological and gene therapy, etc. Among them, the use of radiation therapy is getting more and more attention, and it is changing from the past palliative treatment to current curable treatment. From an oncologic point of view, a narrow margin <1 cm and microvascular invasion is not safe and is often associated with higher rates of recurrence and shorter patient survival.On the other hand, it is also believed that most intrahepatic recurrences arise from multicentric carcinogenesis and are distant from the resection margin. To address this issue, the investigators are going to conduct a series of retrospective and prospective studies to investigate the effect of adjuvant Radiotherapy for centrally located hepatocellular carcinoma after narrow margin (<1 cm) hepatectomy on tumor recurrence.

ELIGIBILITY:
Inclusion Criteria:

1. Patients were pathologically diagnosed as BCLC-A stage hepatocellular carcinomas, liver function were Child-Pugh class A or liver function changed from class B to class A after short-term liver treatment, PS scored 0-1, and accepted hepatocellular carcinomas resection (R0 resection).
2. No recurrence was found within 3-4 weeks after surgery.
3. pathologically confirmed as narrow margin (the closest distance from margin to tumor capsule (<1 cm) and microvascular invasion was found in tumor capsule and adjacent tissues junction (material selection and pathological diagnosis were based on "Standardization pathology Guide of primary liver cancer 2015 edition" ).
4. Postoperative radiotherapy was the only combination therapy within one month after surgery.
5. Radiation range was margin radiation along and/or joint portal vessels radiotherapy.
6. No lymph node and distant metastasis before surgery.

Exclusion Criteria:

1. Patients were pathologically diagnosed as BCLC-B, C, D stage hepatocellular carcinomas, liver function were Child-Pugh class C, PS scored ≥2. Or primary liver cancer patients were pathologically diagnosed as cholangiocarcinoma or mixed type liver cancer. Or patients did not accept hepatectomy.
2. Patients received transcatheter arterial chemoembolization, chemotherapy, targeted medicine or other anti-cancer therapy before surgery.
3. Recurrence was found within 3-4 weeks after surgery.
4. Postoperative adjuvant therapy included treatment other than radiotherapy within one month after surgery.
5. Radiation range involved lymph node other than portal vein area.
6. Lymph node and distant metastasis were diagnosed before surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 620 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-11-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
overall survival | 5years

CONTACTS AND LOCATIONS:
Locations (1):
- TaoBai, Nanning, Guangxi, China